CLINICAL TRIAL: NCT02910401
Title: Clinical Response to Rhinovirus Challenge in Human Asthmatics
Brief Title: Clinical Response to Rhinovirus Challenge
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Larry Borish, MD, Professor of Medicine and Microbiology, University of Virginia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 19157; 1U01AI123337 (NIH)
Record Dates: First submitted 2016-09-08; First posted 2016-09-22 (Estimated); Results first posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Asthma; Allergic Rhinitis
MeSH Terms: conditions — Asthma; Rhinitis, Allergic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Asthmatic (Active Comparator): Asthmatic subjects will be infected with Rhinovirus (GMP RV16 human (H)RV-16)
  Interventions: Biological: Rhinovirus (GMP RV16 HRV-16)
- Allergic rhinitis (Active Comparator): Allergic rhinitis subjects will be infected with Rhinovirus (GMP RV16 HRV-16)
  Interventions: Biological: Rhinovirus (GMP RV16 HRV-16)
- Healthy control (Active Comparator): Healthy controls will be infected with Rhinovirus (GMP RV16 HRV-16)
  Interventions: Biological: Rhinovirus (GMP RV16 HRV-16)

INTERVENTIONS:
Biological: Rhinovirus (GMP RV16 HRV-16) — 300 tissue culture infectious dose (TCID)50 mg/ml intranasal one time only

SUMMARY:
Rhinovirus (RV) infections represent the most common cause of asthma exacerbations in children and adolescents. The investigators hypothesize that the immune responses generated in the nose of allergic rhinitics and asthmatics underlie subsequent systemic modulation of the immune system, and that - in susceptible individuals (i.e., those with pre-existing asthma) - this modified nasal milieu is responsible for the asthma exacerbation.

Open label single center study in asthmatics as well as allergic rhinitis (AR) and healthy controls. All subjects will undergo good manufacturing practice (GMP) RV16 inoculation and responses will be compared between the 3 cohorts.

DETAILED DESCRIPTION:
Primary objectives are:

To determine whether RV increases expression of interleukin (IL)-25 transcripts by nasal epithelial cells in the asthma and AR but not control cohorts at the peak of infection (days 3 and 4).

To determine whether RV increases lower respiratory symptoms in the asthma but not AR and control cohorts.

To determine whether asthmatics and allergic rhinitics will demonstrate an increased severity of infection in comparison to control subjects.

Secondary objectives are:

1. To determine whether asthmatic and AR cohorts demonstrate increased IL-25 transcript expression over the course of RV infection
2. To determine whether asthmatic and AR cohorts demonstrate increased expression of mRNA transcripts of a type 2 cytokine-inducing profile (IL-33 and thymic stromal lymphopoietin (TSLP)).
3. To determine whether increased transcript expression of this type 2 cytokine-inducing profile can be corroborated as increased expression of protein.
4. To determine whether RV infection in the asthma cohort is associated with increases in biomarkers of inflammation.
5. To determine whether increased severity of RV infection in the asthma and AR cohorts will be associated with more symptoms.
6. To determine whether increased severity of RV infection in the asthma and AR cohorts is related to decreased innate immunity.

ELIGIBILITY:
Inclusion Criteria:

All subjects:

1. Subjects must be able to understand and provide written informed consent.
2. Age 18 to ≤40 years of age, any gender, any racial/ethnic origin
3. Female subjects of childbearing potential must have a negative pregnancy test upon study entry (day -7) and before each procedure involving pharmacologic interventions (days 0, 4, and 7).
4. Female (and male) subjects with reproductive potential, must agree to use FDA approved methods of birth control for the duration of the study such as, but not limited to, birth control pills, contraceptive foam, diaphragm, IUD, abstinence, or condoms.
5. Participants must be willing to comply with study procedures and requirements.
6. Negative test for serum neutralizing antibody to RV16 at enrollment visit (<1:8) (Visit 1).

Allergic Rhinitis Subjects:

1. Allergy as determined by ≥1 positive prick skin test (wheal ≥5 mm diameter and 3mm larger than the diluent control) to Virginia inhalant panel within 5 years, and a history of symptoms of sneezing, rhinorrhea, pruritus, nasal congestion, and/or allergic conjunctivitis on natural exposure to relevant allergens.
2. Negative methacholine challenge (less than 20% decline in functional expiratory volume in 1 second (FEV1) at ≤8mg/ml) within 1 year
3. FEV1 ≥80% predicted, FEV1/FVC ≥80%.
4. No history of wheezing with viral infection in the last 6 years, and no use of rescue inhalers or long-term controllers for asthma in the last 6 years.

Allergic Asthmatic Subjects:

1. Allergy as determined by ≥1 positive prick skin test (wheal ≥5 mm diameter and 3mm larger than the diluent control) to Virginia inhalant panel. Subjects are not required to have allergy symptoms at the time of study. Subjects will report history of symptoms of sneezing, rhinorrhea, pruritus, nasal congestion, and/or allergic conjunctivitis on natural exposure to relevant allergens.
2. Asthma determined by physician diagnosis and by a positive methacholine challenge (at least 20% fall in FEV1 at a methacholine concentration of ≤8 mg/ml) at screening protocol visit before enrollment (obtained within the past year).
3. Asthma must be controlled as determined by asthma control test (ACT) score ≥20 and normal lung function (FEV1>70% predicted or FEV1/FVC ratio >75% for subjects with FVC values between 80 and 87% predicted whose FEV1 values fall below 70%) at Visits 1 and 2.

Exclusion Criteria:

1. Positive test for serum neutralizing antibody to RV16 at enrollment visit (≥1:8) (Visit 1).
2. Upper airway modified Jackson criteria symptom scores ≥7 at time of inoculation.
3. Chronic heart disease including bradycardia, lung diseases other than asthma, or other chronic illnesses including epilepsy, peptic ulcer disease, thyroid disease, urinary tract infection, vagotonia, autoimmune disease, primary or secondary immunodeficiency or any household contacts who are known to be immune deficient. Any medical conditions that could be adversely affected by the administration of cholinergic agent.
4. Any use of corticosteroids, leukotriene (LT) modifiers, antihistamines, omalizumab, theophylline, long-acting anti-muscarinic antagonists (LAMAs), long-acting beta-agonists (LABAs), nedocromil, cromolyn use on a daily basis within 4 weeks prior to Visit 1.
5. Current use of ß-blockers or cholinesterase inhibitors (for myasthenia gravis).
6. ß2-agonist use ≥4 days/week in any week or ≥2 nights/month during the month before Visit 1.
7. Recent (within 1-yr) asthma exacerbation requiring urgent care visit (unless the treatment involved only the use of a bronchodilator), hospitalization, or oral CCS
8. Intubation or management in the intensive care unit (ICU) for an asthma exacerbation ever.
9. An upper or lower respiratory tract infection within 2 months prior to enrollment.
10. Previous nasal or sinus surgery within the last 12 months
11. >5 pack-year smoking history or any smoking within the past 6 mos.
12. Hemoglobin <11.5 g/dL for non-African American subjects or hemoglobin < 11.0 g/dL for African American subjects detected at Visit 1.
13. Laboratory values (other than hemoglobin and absolute neutrophil count (ANC)) measured at Visit 1 that are considered to be of clinical relevance by the Investigator.
14. Absolute neutrophil count (ANC) <1500 cells/mm3 (or 1.5 K/µL) or absolute lymphocyte count (ALC) <800 cells/mm3 detected at Visit 1.
15. Use of investigational drugs within 12 weeks of participation
16. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2022-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry Borish, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Feng X, Lawrence MG, Payne SC, Mattos J, Etter E, Negri JA, Murphy D, Kennedy JL, Steinke JW, Borish L. Lower viral loads in subjects with rhinovirus-challenged allergy despite reduced innate immunity. Ann Allergy Asthma Immunol. 2022 Apr;128(4):414-422.e2. doi: 10.1016/j.anai.2022.01.007. Epub 2022 Jan 12. PMID 35031416

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Asthmatic | Allergic Rhinitis | Healthy Control
Started | 6 | 17 | 15
Completed | 5 | 17 | 13
Not Completed | 1 | 0 | 2
Not completed — Study closure Study closure | 0 | 0 | 2
Not completed — Physician Decision | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Asthmatic | Allergic Rhinitis | Healthy Control | Total
Number analyzed (Participants) | 6 | 17 | 15 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 17 | 15 | 38
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.7 (0.5) | 21.5 (0.7) | 22.8 (0.4) | 21.9 (0.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 10 | 8 | 21
  Male | 3 | 7 | 7 | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 6 | 17 | 15 | 38

OUTCOME MEASURES:

1. Primary Outcome: Change in Symptom Scores Induced by the Rhinovirus Using Jackson Criteria Including Nasal Congestion, Drainage, Cough, Wheezing
Description: Jackson criteria subjective score for: nasal secretion (0 - none; 1 - mild; 2 - moderate; 3 - severe), congestion (0 - none; 1 - mild; 2 - moderate; 3 - severe), cough (0 - none; 1 - mild; 2 - moderate; 3 - severe), pain/pressure (0 - none; 1 - mild; 2 - moderate; 3 - severe). Scoring was done twice a day and total score reported for a maximum range for each day of 0-24. Scoring was done daily for 4 weeks.
Time Frame: Change in symptom score from day 0 to day 4 after inoculation with the rhinovirus
Population: Jackson symptom score
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Asthmatic | Allergic Rhinitis | Healthy Control
Number analyzed (Participants) | 5 | 17 | 13
score on a scale | 5.0 [0 to 10] | 4.2 [0 to 10] | 2.8 [0 to 10]

ADVERSE EVENTS:
Time Frame: Adverse events were reported for each individual from the time of signing the informed consent form through the end of visit safety visit which was 4 weeks after the viral inoculation (5 weeks after signing consent form). All AEs were recorded on a log for the duration of the study (5 years).
Arm/Group | Asthmatic | Allergic Rhinitis | Healthy Control
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/17 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/17 | 0/15
Other Adverse Events (participants affected / at risk) | 0/6 | 1/17 | 0/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Asthmatic (N=6) | Allergic Rhinitis (N=17) | Healthy Control (N=15)
Abdominal pain (Gastrointestinal disorders) | NA | 1 | NA — Stomach ache

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-04): https://cdn.clinicaltrials.gov/large-docs/01/NCT02910401/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-09): https://cdn.clinicaltrials.gov/large-docs/01/NCT02910401/ICF_001.pdf